CLINICAL TRIAL: NCT05082584
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Once Daily Oral Vadadustat for The Treatment of Pediatric Subjects With Anemia of Chronic Kidney Disease Naive to Erythropoiesis-stimulating Agents
Brief Title: Study to Evaluate the Safety and Efficacy of Oral Vadadustat in Pediatric Participants With Anemia of Chronic Kidney Disease Naive to Erythropoiesis-Stimulating Agents
Acronym: CORRECTION
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0042
Record Dates: First submitted 2021-09-28; First posted 2021-10-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: anemia; chronic kidney disease; erythropoiesis stimulating agent; dialysis; vadadustat; pediatric population; children; kidney disease; hypoxia-inducible factor (HIF) prolyl hydroxylase inhibitor
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Diseases | interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vadadustat (Experimental): Cohort 1: participants with ≥12 years to <17 years; Cohort 2: participants with ≥6 years to <12 years; Cohort 3(a): participants with ≥2 years to <6 years; and Cohort 3(b): participants with ≥4 months to <2 years
  Interventions: Drug: Vadadustat

INTERVENTIONS:
Drug: Vadadustat — Vadadustat tablet orally once a day for 52 weeks
  Other Names: AKB-6548

SUMMARY:
This study will assess the safety and efficacy of once daily dosing of vadadustat for the treatment of pediatric participants with anemia of chronic kidney disease (CKD) naive to erythropoiesis-stimulating agent (ESA) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anemia of chronic kidney disease (CKD)
* Diagnosis of non-dialysis-dependent (NDD) CKD with an estimated glomerular filtration rate of greater than (>) 10 and less than (<) 60 milliliters/minute/1.73 meters^2 (mL/min/1.73 m^2 ) or diagnosis of dialysis dependent (DD) CKD
* Mean screening hemoglobin (Hb) <10.0 grams/deciliters (g/dL)
* Transferrin Saturation ≥ 20%

Exclusion Criteria:

* Anemia due to a cause other than CKD
* Active bleeding or recent clinically significant blood loss
* Treatment with an erythropoiesis-stimulating agents (ESA) within 8 weeks prior to Screening
* History of sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red Blood Cells transfusion within 4 weeks
* Serum albumin level <2.5 g/dL
* Uncontrolled hypertension
* Active malignancy or treatment for malignancy within the past 2 years prior to Screening
* Evidence of iron overload or diagnosis of hemochromatosis
* Known hypersensitivity to vadadustat or any excipients in vadadustat tablet

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Hemoglobin (Hb) Values Between Baseline and the Primary Evaluation Period (Average Hb From Weeks 21 to 28) | Baseline; Weeks 21 to 28

SECONDARY OUTCOMES:
Time to Achieve First Hb Levels ≥10.0 grams/deciliters (g/dL) | Up to Week 52
Number of Participants With Mean Hb Values Within the Target Range During the Primary Evaluation Period | From Week 21 to Week 28
Number of Participants With Mean Hb Values Within the Target Range During the Extension Period | From Week 29 to Week 52
Number of Participants With Treatment-emergent Adverse Events and who Discontinued From the Study due to Adverse Events | Up to Week 56
Maximum Observed Plasma Concentration (Cmax) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC 0-t) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Time to Reach Cmax (Tmax) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Terminal Elimination Half-Life (t1/2) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Serum Erythropoietin (EPO) | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Reticulocyte Count | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Hb levels | Pre-dose and post-dose at intermediate time points up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (1):
- Research Site, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No